CLINICAL TRIAL: NCT03531151
Title: Magnetic Resonance Imaging of Myocardial Infarction
Brief Title: MRI of Myocardial Infarction
Acronym: MRIMI
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 827697
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction; Myocardial Ischemia; Myocardial Injury; Myocardial Fibrosis; Myocardial Reperfusion Injury; Myocardial Edema; Myocardial Necrosis; Heart Failure; Ischemic Heart Disease; Ischemic Cardiomyopathy; Hemorrhage
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Myocardial Reperfusion Injury; Heart Failure; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) is an enormous health burden affecting approximately 5.1 million people in the US and is the cause of 250,000 deaths each year. Approximately 50% of HF is caused by myocardial ischemia and requires immediate restoration of coronary blood flow to the affected myocardium. However, the success of reperfusion is partly limited by intramyocardial hemorrhage, which is the deposition of intravascular material into the myocardium. Hemorrhagic reperfusion injury has high prevalence and patients have a much greater risk of adverse left ventricular remodeling, risk of fatal arrhythmia, impaired systolic function and are hospitalized at a greater rate. Recent magnetic resonance imaging techniques have improved assessment of reperfusion injury, however, the association between MRI contrasts and reperfusion injury is highly unclear, and lacks specificity to IMH. Improved imaging of IMH and accurate knowledge about its spatial and temporal evolution may be essential for delivery of optimal medical therapy in patients and critical to identify patients most at risk for adverse ventricular remodeling. The overall goal is to investigate the magnetic properties of hemorrhage and develop MRI techniques with improved specificity to hemorrhage. New MRI techniques permit noninvasive assessment of the magnetic susceptibility of tissues and can target tissue iron. Therefore, the investigators hypothesize that MRI imaging of myocardial magnetic susceptibility can map hemorrhagic myocardium. The investigators will perform a longitudinal observational study in patients after reperfusion injury to validate these methods, compare the methods with conventional MR contrasts and develop MR methods for imaging humans.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 80
* Patients must be able to read and understand English
* Participants must sign the informed consent form
* Elevated and delayed peak creatine kinase-MB and troponin I (cTnI) and troponin T (cTnT) in blood serum,
* ST elevation detected on ECG

Exclusion Criteria:

* contraindications to cardiac MRI, including claustrophobia
* advanced renal disease (estimated glomerular filtration rate 30 mL/min) or hypersensitivity to gadolinium
* presence of a cardiac pacemaker or implanted cardiac cardioverter defibrillator
* pregnancy
* personal or family history of hypertrophic cardiomyopathy
* inability to provide informed consent
* history of seizure disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population specific to this project are ST-elevated myocardial infarction (STEMI) patients being treated with reperfusion therapy.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
ejection fraction | <36 hours to >6 months

SECONDARY OUTCOMES:
relaxation times | <36 hours to >6 months
extracellular volume fraction | <36 hours to >6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided